CLINICAL TRIAL: NCT07174115
Title: A Phase IIa Clinical Study to Evaluate the Efficacy and Safety of HTMC0658 Tablets in the Treatment of Chronic Rhinosinusitis Without Nasal Polyps
Brief Title: A Study to Evaluate the Efficacy and Safety of HTMC0658 Tablets in the Treatment of Chronic Rhinosinusitis Without Nasal Polyps
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yidian Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PY-HTMC0658-IIa-01
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Sinusitis Without Nasal Polyps
Keywords: chronic sinusitis without nasal polyps; Dipeptidyl peptidase 1; neutrophil-related inflammatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HTMC0658 (Experimental): Participants will receive HTMC0658 tablet, orally, QD for 12 weeks along with mometasone furoate nasal spray (MFNS) by nasal route as background therapy at a stable dose according to the Investigator's discretion and local guidance.
  Interventions: Drug: HTMC0658

INTERVENTIONS:
Drug: HTMC0658 — HTMC0658 tablet
  Other Names: YD0293 tablet

SUMMARY:
The purpose of this clinical trial is to assess the efficacy and safety of HTMC0658 tablets in treating subjects with chronic rhinosinusitis without nasal polyps (CRSsNP).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 75 years, inclusive, of either sex.
2. Body Mass Index (BMI) calculated as weight in kilograms divided by the square of height in meters (kg/m²), with a BMI of at least 18.5.
3. Subjects must meet the diagnostic criteria for chronic rhinosinusitis as defined in the "Chinese Chronic Rhinosinusitis Diagnosis and Treatment Guidelines (2024)," with a disease duration exceeding 12 weeks.
4. During the screening period, nasal endoscopy must reveal bilateral pathological changes in the nasal mucosa, such as edema and purulent discharge, or a CT scan must show bilateral sinus involvement.
5. During the screening period, a CT scan must demonstrate bilateral sinus involvement, with at least one sinus on each side scoring ≥ 1 point on the Lund-MacKay (LMK) scale.
6. During the screening period, the Nasal Congestion Score (NCS) must be ≥ 2 points.
7. During the screening period, the Composite Symptom Score (CSS) for nasal congestion, rhinorrhea, and facial pain/pressure must be ≥ 5 points.
8. During the screening period, the Sino-Nasal Outcome Test-22 (SNOT-22) total score must be ≥ 20 points.
9. Subjects must have been on a stable daily dose of mometasone furoate nasal spray (MFNS) for at least 4 weeks prior to enrollment.
10. Subjects with asthma or chronic obstructive pulmonary disease (COPD) must have had stable conditions without exacerbations in the 3 months prior to screening (e.g., no emergency room visits, hospitalizations, or systemic corticosteroid use). The use of inhaled corticosteroids must have been at a stable dose, with continuous use for at least 3 months prior to screening, and planned continuation throughout the study period.
11. Subjects must fully understand the purpose, nature, methodology, and potential adverse events of the trial, voluntarily participate in the trial, and provide written informed consent, or have an authorized legal representative provide informed consent.

Exclusion Criteria:

1. Presence of nasal polyps confirmed by nasal endoscopy during the screening period, or a history of nasal polyps.
2. Requirement for systemic corticosteroids as maintenance therapy during the screening period.
3. Diagnosis of cystic fibrosis (CF) or primary ciliary dyskinesia.
4. Undergone nasal surgery within 4 weeks prior to screening, or scheduled for sinus surgery during the study period.
5. Presence of significant craniofacial structural abnormalities or severe nasal septal deviation.
6. Radiological suspicion or confirmed diagnosis of invasive fungal rhinosinusitis, odontogenic sinusitis, osteoma, or nasal tumor.
7. Presence of a disease or comorbidity that would interfere with the assessment of the primary efficacy endpoints (e.g., subjects with seasonal allergic rhinitis whose symptoms coincide with the study treatment period; subjects with moderate to severe atopic dermatitis requiring treatment with potent topical corticosteroids, topical calcineurin inhibitors, or biologics; subjects with acute upper respiratory tract infection that, in the investigator's judgment, would affect nasal symptom scoring).
8. Presence of an acute infection requiring antibiotic treatment within 4 weeks prior to screening.
9. Inflammatory or autoimmune diseases requiring systemic biologic therapy or immunosuppressive agents (including but not limited to immunodeficiency diseases).
10. Known allergy or intolerance to any component of the investigational medicinal product or background therapy.
11. Subjects with a past or current diagnosis of periodontitis or palmoplantar keratoderma due to functional deficiency of dipeptidyl peptidase 1 (DPP1), or the presence of the following at screening:a. Subjects with current signs of gingivitis/periodontitis.b. Subjects with a history of palmoplantar keratoderma or erythema.
12. Receipt of drugs that may cause skin hyperkeratosis (e.g., tumor necrosis factor-α antagonists) within 4 weeks prior to screening.
13. Patients who have used strong CYP3A4 or CYP2D6 inhibitors or inducers within 14 days prior to the first administration of the investigational medicinal product.
14. Subjects with elevated liver function test results during the screening period and currently requiring treatment for liver disease. Elevated liver function tests are defined as: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 × upper limit of normal (ULN), or total bilirubin (TBIL) > 1.5 × ULN.
15. Subjects with positive test results for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, and/or syphilis serology during the screening period.
16. Current smokers (defined as adults who have smoked at least 100 cigarettes in their lifetime and are currently smoking) or those who cannot abstain from smoking during the trial.
17. Subjects who have participated in other drug or medical device trials within 3 months prior to the start of this trial or are currently enrolled in another clinical trial.
18. Male subjects who plan to donate sperm or have a fathering plan from the start of dosing until 90 days after the last dose and are unwilling to use effective non-pharmacological contraceptive measures.
19. Female subjects who plan to donate oocytes or have a pregnancy plan from the start of dosing until 30 days after the last dose and are unwilling to use effective non-pharmacological contraceptive measures.
20. Pregnant or breastfeeding women.
21. Subjects whom the investigator deems unsuitable for participation in this study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Lund-MacKay (LMK) score on sinus CT scan at Week 12 | Baseline to 12 weeks
  Lund-MacKay (LMK) score for CT scan of the sinuses: This score evaluates the left and right maxillary sinuses, anterior ethmoid sinuses, posterior ethmoid sinuses, sphenoid sinuses, frontal sinuses, and the ostiomeatal complex. Scoring criteria are as follows: For the sinuses: 0 = no abnormality, 1 = partially opacified, 2 = completely opacified; For the ostiomeatal complex: 0 = no obstruction, 2 = obstruction. The score for each side ranges from 0 to 12, with a total possible score of 0 to 24.

SECONDARY OUTCOMES:
Change from baseline in Composite Symptom Score (CSS) at Weeks 4, 8, and 12 | baseline to 4, 8 and 12 weeks
  Composite Symptom Score (CSS) for Chronic Rhinosinusitis: These symptoms are categorized into three types: nasal congestion, facial pain/pressure, and nasal discharge. The scoring criteria are as follows: 0 = no symptoms (absence of noticeable signs or symptoms), 1 = mild symptoms (presence of signs or symptoms that are mild and tolerable), 2 = moderate symptoms (signs or symptoms that are noticeable and uncomfortable but tolerable), 3 = severe symptoms (signs or symptoms that are intolerable and interfere with daily activities and/or sleep). The total score ranges from 0 to 9.
Change from baseline in the Sino-Nasal Outcome Test-22 (SNOT-22) scale score at Weeks 4, 8, and 12 | baseline to 4, 8, and 12 weeks
  The SNOT-22 is a subject-completed questionnaire that consists of 22 symptoms and social/emotional consequences of their nasal disorder across several domains including: rhinologic, extra-nasal rhinologic, ear/facial pain, psychological dysfunction, and sleep dysfunction. Total scores range from 0-110. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be, and total scores are calculated by adding scores together.
Change from baseline in the Visual Analog Scale (VAS) score for the severity of rhinosinusitis at Weeks 4, 8, and 12 | baseline to 4, 8, and 12 weeks
  Visual Analogue Scale (VAS) for the Severity of Chronic Rhinosinusitis: Draw a 10 cm straight line on a piece of white paper. Label one end as "No Disturbance" and the other end as "The Worst Disturbance That Can Be Imagined" to create the VAS. The subject marks a point on the line corresponding to the severity of their sinusitis symptoms. The distance from the starting point to the marked point represents the quantified severity of the symptoms.
Change from baseline in Nasal Congestion Score (NCS) at Weeks 4, 8, and 12 | baseline to 4, 8, and 12 weeks
  Nasal Congestion Score: The scoring criteria are as follows: 0 = No symptoms (no obvious signs/symptoms), 1 = Mild symptoms (signs/symptoms exist but are mild and tolerable), 2 = Moderate symptoms (signs/symptoms are obvious, causing discomfort but still tolerable), 3 = Severe symptoms (signs/symptoms are unbearable, affecting daily activities and/or sleep). The total score ranges from 0 to 3.
Patient Global Impression of Change (PGIC) scale score at Week 12 | 12 weeks
  The global impression of change will be assessed using a subject-completed PGIC scale, which ranges from 1 to 7: 1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse.
Proportion of subjects requiring rescue therapy (antibiotics, systemic corticosteroids, and/or nasal surgery) due to worsening of any chronic rhinosinusitis symptoms within 12 weeks. | 12 weeks
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | baseline to 16 weeks
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs), as well as changes in vital signs and laboratory test results, etc.
Plasma Concentration of HTMC0658 | Pre-dose and at multiple timepoints post-dose up to Day 30
Changes in serum neutrophil elastase (NE) concentration | Baseline to 4, 8, and 12 weeks
  Changes from baseline in serum neutrophil elastase (NE) concentration at Weeks 4, 8, and 12 of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Luoyang First People's Hospital, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No